CLINICAL TRIAL: NCT00310232
Title: Randomized Trial of Epoetin Alfa in Patients With Advanced Non-Small Cell Carcinoma of the Lung (EPO-CAN-20)
Brief Title: Epoetin Alfa in Advanced Non-Small Cell Lung Cancer (EPO-CAN-20)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Recommendation of DSMB for safety issue, increased mortality with study drug.
Sponsor: Ontario Clinical Oncology Group (OCOG) (Other)
Collaborators: Ortho Biotech, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CTA-Control-076080; HC File 9427-J0921-22C
Record Dates: First submitted 2006-03-31; First posted 2006-04-03 (Estimated); Last update posted 2024-04-02 (Actual); Status verified 2024-04

CONDITIONS: Non-Small-Cell Lung Carcinoma; Lung Cancer; Anemia
Keywords: Quality of Life; Blood transfusion
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms; Anemia | interventions — Epoetin Alfa

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Epoetin Alfa

SUMMARY:
The general objective of this study is to improve the Quality of Life (QoL) of selected patients with advanced carcinoma of the lung. The specific objective is to evaluate the effect of treatment with epoetin alfa (recombinant human erythropoietin) on anemia related QoL and anemia in non-small cell lung cancer patients with advanced stage disease and underlying anemia of malignancy.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed non-small cell lung cancer (squamous cell, large cell, adenocarcinoma, or some combination of these), with clinical or pathological stage III or IV, or recurrent disease; and
2. Hemoglobin level at or below 120 g/L; and
3. At least 18 years of age;

Exclusion Criteria:

1. Systemic platinum-based chemotherapy for lung cancer during the previous two months or planned platinum-based chemotherapy within the next three months;
2. Patients previously treated with high dose thoracic radiation (>10 fractions), or surgery, without objective evidence of disease recurrence;
3. Planned high dose thoracic radiation therapy (>10 fractions);
4. A clinically active malignancy, other than the underlying lung cancer which is expected to influence QoL;
5. Expected survival of three months or less;
6. ECOG Performance status of 3 or 4 (see Appendix D);
7. Multiple CNS metastasis or a single CNS lesion that does not demonstrate radiographic stability (Screening CT of head required only if symptomatic, no radiographic follow-up of single resected lesions required);
8. Blood transfusions within the last 14 days;
9. Previous use of erythropoietin;
10. Anemia due to factors other than cancer / radiotherapy (e.g. hemolysis or gastrointestinal bleeding);
11. Evidence of untreated folate or vitamin B12 deficiency;
12. History of uncontrolled hypertension or diastolic blood pressure greater than 100 mm Hg;
13. History of seizure disorder;
14. Known hypersensitivity to mammalian cell-derived products, albumin or any component of the study drug;
15. Pregnancy, lactation or parturition within the previous 30 days;
16. Unwillingness or inability to complete the required QoL questionnaires;
17. Mental incompetence, including psychiatric or addictive disorders which would preclude meaningful completion of questionnaires;
18. Geographically inaccessible for treatment or follow-up evaluations;
19. Currently enrolled in an ongoing therapeutic study;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2001-02; Study Completion 2004-04 (Actual)

PRIMARY OUTCOMES:
Change in anemia and fatigue related QoL at 12 weeks following randomization | 12 weeks following randomization

SECONDARY OUTCOMES:
Overall QoL and domain-specific QoL scores | 16 weeks following randomization
hemoglobin and hematocrit levels | 6 months from randomization
number of transfusions | 6 months from randomization

CONTACTS AND LOCATIONS:
Overall Officials: Jim Wright, MD, Study Chair — Hamilton Regional Cancer Centre; Mark Levine, MD, Study Director — Ontarion Clinical Oncology Group
Locations (15):
- Canada (15):
  - Tom Baker Cancer Centre, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - Cancer Care Manitoba, Winnipeg, Manitoba
  - St. John Regional Hospital, Saint John, New Brunswick
  - Newfoundland Cancer Treatment & Research Foundation, St. John's, Newfoundland and Labrador
  - Nova Scotia Cancer Centre, Halifax, Nova Scotia
  - Northeastern Ontario Regional Cancer Centre, Greater Sudbury, Ontario
  - Hamilton Regional Cancer Centre (Juravinski), Hamilton, Ontario
  - London Regional Cancer Centre, London, Ontario
  - Hotel Dieu Hospital, Saint Catherines, Ontario
  - Toronto East General Hospital, Toronto, Ontario
  - Toronto Sunnybrook Regional Cancer Centre, Toronto, Ontario
  - Princess Margaret Hospital, Toronto, Ontario
  - Windsor Regional Cancer Centre, Windsor, Ontario
  - McGill University Clinical Trials Operations, Montreal, Quebec

REFERENCES:
- [Result] Wright JR, Ung YC, Julian JA, Pritchard KI, Whelan TJ, Smith C, Szechtman B, Roa W, Mulroy L, Rudinskas L, Gagnon B, Okawara GS, Levine MN. Randomized, double-blind, placebo-controlled trial of erythropoietin in non-small-cell lung cancer with disease-related anemia. J Clin Oncol. 2007 Mar 20;25(9):1027-32. doi: 10.1200/JCO.2006.07.1514. Epub 2007 Feb 20. PMID 17312332